CLINICAL TRIAL: NCT03704506
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial of the Efficacy and Safety of Treating Acute Tonsillitis With Reyanning Mixture Alone/in Combination With Antibiotics.
Brief Title: Registration of the Study of Reyanning Mixture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Beijing Chao Yang Hospital (Other); Wangjing Hospital, China Academy of Chinese Medical Sciences (Other); Beijing First Hospital of integrated Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reyanning mixture
Record Dates: First submitted 2018-10-07; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Acute Tonsillitis
Keywords: Reyanning mixture; efficacy; safety; randomized; double-blind; placebo-controlled; multicenter; antibiotics
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treatment group 1 (Experimental): Reyanning mixture+amoxil capsule simulator
  Interventions: Drug: Reyanning mixture; Drug: amoxil capsule simulator
- treatment group 2 (Experimental): Reyanning mixture +amoxil capsule
  Interventions: Drug: Reyanning mixture; Drug: amoxil capsule
- control group (Active Comparator): Reyanning mixture simulator +amoxil capsule
  Interventions: Drug: amoxil capsule; Drug: Reyanning mixture simulator

INTERVENTIONS:
Drug: Reyanning mixture — Reyanning mixture , 20ml by mouth , 3 times per day for 7 days
  Other Names: Reyanning
  Arms: treatment group 1; treatment group 2
Drug: amoxil capsule — amoxil capsule , 0.5g by mouth , 3 times per day for 7 days
  Other Names: amoxicillin
  Arms: control group; treatment group 2
Drug: Reyanning mixture simulator — Reyanning mixture simulator , 20ml by mouth , 3 times per day for 7 days
  Other Names: Reyanning simulator
  Arms: control group
Drug: amoxil capsule simulator — amoxil capsule simulator , 0.5g by mouth , 3 times per day for 7 days
  Other Names: amoxicillin simulator
  Arms: treatment group 1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of treating with acute tonsillitis using Reyanning mixture alone/in combination with antibiotics, and its function of reducing the use of antibiotics.

DETAILED DESCRIPTION:
In order to evaluate the efficacy,safety and the function of reducing the use of antibiotics of Reyanning mixture (a mixture of Chinese herbal medicine) in treating with acute tonsillitis, a randomized, double-blind, placebo-controlled, multicenter clinical trials will be established. According to the relevant regulations of the China Food and Drug Administration(CFDA), 144 cases need to be registered at least. The aim population is who suffering of acute tonsillitis from October 2018 to December 2019.These cases will be randomly divided into treatment group 1(Reyanning mixture +amoxil capsule simulator),treatment group 2(Reyanning mixture +amoxil capsule) and control group(Reyanning mixture simulator +amoxil capsule).Each group will be treated for 7 days and followed up for 3 times . The main indicators include the recovery time/rate and antibiotic duration/dosage. And the vanish rate of single symptom/physical sign, the ratio of white blood cell count(WBC) recovery, the time of fever will be observed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of acute tonsillitis;
2. Meet the traditional Chinese medicine symptom diagnostic criteria of external wind-heat type and excessive heat in the lung and stomach type;
3. 18 years≤age≤65 years;
4. course of disease within 72 hours;
5. sign informed consent.

Exclusion Criteria:

1. common cold,influenza, acute laryngopharyngitis, pharyngeal diphtheria, wensang's isthmitis.
2. complicated with acute tracheobronchitis,pneumonia,rheumatic fever, acute glomerulonephritis or rheumatic heart disease.
3. complicated with severe angiocardiopathy, cerebrovascular disease, hemopoietic system disease or psychopath.
4. liver or kidney function is abnormal(ALT>1.5 times upper limit of normal; Cr>upper limit of normal); diabetic.
5. WBC<10×109/L and neutrophilic granulocyte percentage<75%;or WBC ≥20×109/L;
6. gestational, lactating women or who planning to get pregnant within half a year.
7. already accept similar traditional Chinese medicine or antibiotic within 48 hours before registered.
8. joining other clinical trials or allergic to any drug in this trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-10-22 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
recovery time | after 3 days of medication
  The recovery time will be observed. Recovery means that the main signs and symptoms score is zero, and body temperature is below 37.3 ℃ maintaining for at least 24 hours.
recovery time | after 7 days of medication
  The recovery time will be observed. Recovery means that the main signs and symptoms score is zero, and body temperature is below 37.3 ℃ maintaining for at least 24 hours.
recovery rate | after 3 days of medication
  The recovery rate will be observed. Recovery means that the main signs and symptoms score is zero, and body temperature is below 37.3 ℃ maintaining for at least 24 hours.
recovery rate | after 7 days of medication
  The recovery rate will be observed. Recovery means that the main signs and symptoms score is zero, and body temperature is below 37.3 ℃ maintaining for at least 24 hours.
antibiotic duration | after 7 days of medication
  The duration of antibiotic will be observed.
antibiotic dosage | after 7 days of medication
  The dosage of antibiotic will be observed.

SECONDARY OUTCOMES:
the vanish rate of single symptom/physical sign | after 3 days of medication
  The single symptom/physical sign include tonsil redness, pharyngeal pain, and fever.
the vanish rate of single symptom/physical sign | after 7 days of medication
  The single symptom/physical sign include tonsil redness, pharyngeal pain, and fever.
the ratio of WBC recovery | after 7 days of medication
  The ratio of WBC recovery refers to the percentage of white blood cell count which return to normal range after 7 days of medication.
the time of fever relieving | after 7 days of medication
  The time of fever relieving means that the duration from the first medication to the body temperature drops below 37.3℃ maintaining for at least 24 hours.

OTHER OUTCOMES:
To observe if Reyanning mixture causes liver function damage. | after 7 days of medication
  to assess the liver function indicators
To observer if Reyanning mixture impacts renal function | after 7 days of medication
  to assess the renal function indicators ,including serum creatinine(Cr) and glomerular filtration rate( eGFR)
To observer if Reyanning mixture causes renal damage | after 7 days of medication
  to assess the urinalysis indicators

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No